CLINICAL TRIAL: NCT02570269
Title: Prospective Randomized Comparison Between a Flexible Fiberoptic Intubation Via the Ambu® Aura Gain™ Airway and the Slotted Guedel Tubus in Terms of Time to a Completed Airway Management and Patient Safety.
Brief Title: Prospective Comparison of Oral Intubation Via - Ambu® Aura Gain™ vs Slotted Guedel Tubus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Responsible Party: Principal Investigator, Berthold Moser, Principal Investigator, Schulthess Klinik
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Schulthess_Anä_6
Record Dates: First submitted 2015-09-23; First posted 2015-10-07 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2016-04

CONDITIONS: Adverse Anesthesia Outcome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AuraGain (Active Comparator): The patient will get a fiberoptic Intubation via the AuraGain larynxmask
  Interventions: Procedure: AuraGain
- Slotted Guedeltubus (Placebo Comparator): The patient will get a fiberoptic intubation via the slotted Guedeltubus
  Interventions: Procedure: Slotted Guedeltubus

INTERVENTIONS:
Procedure: AuraGain — Fiberoptic Intubation
  Arms: AuraGain
Procedure: Slotted Guedeltubus — Fiberoptic Intubation
  Arms: Slotted Guedeltubus

SUMMARY:
The study has to show that an intubation with the AuraGain Laryngeal mask could bring the same benefits in terms of intubation in clinical practice, as the slotted Guedel tubus.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18
* ASA 1 -2
* Surgery of the shoulder, elbow, hand, hip, knee or foot
* Signed consent form

Exclusion Criteria:

* Patients with expected difficulties regarding to the intubation
* Patients with diseases / anatomical changes in the area of the pharynx, the larynx, the trachea, the esophagus or the stomach
* Not sober
* Increased risk of aspiration
* BMI > 35 kg/m2
* Acute disease which could affect the suitability of the anesthesia
* Patients in which the use of a laryngeal mask is contraindicated or otherwise not possible
* Patients with a disease which prevents an accurate examination of the patients (eg neuromuscular, mentally, metabolic disease)
* Drug abuse in the recent past
* Legal incompetence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Intubation time | Intraoperative
  Time to complete the Intubation in seconds

SECONDARY OUTCOMES:
Intubation attempts | Intraoperative
  The number of intubation attempts will be recorded (eg 1, 2, 3...)
Esophagal Intubation attempts | Intraoperative
  The number of esophagal intubation attempts will be recorded (eg 1, 2, 3...)
Resistance measurement of the Insertion as assessed by a four point scoring system | Intraoperative
  1/2/3/4
Position of the mask as assessed by the Brimacombe Score | Intraoperative
  4/3/2/1
Pain after Intubation as assessed by a Numeric Rating Scale | Intraoperative/2h postoperative/24h postoperative
  mild/moderate/severe
AE/Complications | Intraoperative/postoperative until 24h
  Occuring AE/Complications will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Moser, MD, Principal Investigator — Schulthess Klinik
Locations (1):
- Schulthess Klinik, Zurich, Switzerland

REFERENCES:
- [Derived] Moser B, Audige L, Keller C, Brimacombe J, Gasteiger L, Bruppacher HR. Flexible bronchoscopic intubation through the AuraGain laryngeal mask versus a slit Guedel tube: a non-inferiority randomized-controlled trial. Can J Anaesth. 2017 Nov;64(11):1119-1128. doi: 10.1007/s12630-017-0936-7. Epub 2017 Jul 17. PMID 28718101